CLINICAL TRIAL: NCT04995913
Title: Development and Evaluation of the Effectiveness of an Online Cognitive Behavioral Intervention Program for Hong Kong People With Social Anxiety Disorder
Brief Title: Online Cognitive Behavioral Intervention Program for Hong Kong People With Social Anxiety Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Research Grants Council, Hong Kong (Other); Stockholm University (Other); Richmond Fellowship Hong Kong (Unknown); Caritas Wellness Link - Tsuen Was (Unknown)
Responsible Party: Principal Investigator, Jiayan Pan, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R2018-18
Record Dates: First submitted 2021-08-06; First posted 2021-08-09 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computer-based (PC) online CBT program (Web version of the EASE Online Program) (Experimental): The Web version of the EASE Online Program delivers the online CBT program through the Program website. It includes 9 online modules, 3 face-to-face/online/telephone counseling sessions, and 2 sessions of virtual reality exposure therapy.
  Interventions: Other: Online cognitive behavioral therapy
- Smartphone-based (App) online CBT program (App version of the EASE Online Program) (Experimental): The App version of the EASE Online Program delivers the online CBT program through a smartphone application. The program content and system functions are the same as those of the Web version.
  Interventions: Other: Online cognitive behavioral therapy
- Waitlist control group (Other): The Waitlist control group will receive the service of the Web version of the EASE Online Program after the two experimental groups completed the service.
  Interventions: Other: Online cognitive behavioral therapy

INTERVENTIONS:
Other: Online cognitive behavioral therapy — The intervention includes 9 online modules, 3 face-to-face/online/telephone counseling sessions, and 2 sessions of virtual reality exposure therapy. Participants will learn and practice a variety of the cognitive behavioral skills to cope with their social anxiety. The functions of the EASE Online Program include animation briefing and debriefing, case demonstration videos, assignment and feedback, forum, internal messaging, reminder, online assessment, online booking and progress checking. The duration of the intervention is 14 weeks.

SUMMARY:
This study developed an online counseling program called "EASE Online" for Hong Kong people with social anxiety disorder. The program effectiveness was evaluated by a randomized controlled trial in reducing social anxiety and improving quality of life of the participants. The 3- and 6-month maintenance effects were also tested.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD), also known as social phobia, is one of the most common mental disorders worldwide. In Hong Kong, the 12-month prevalence of SAD is 3.2% (Lee, Lee & Kwok, 2005) with more than 230,000 sufferers. However, only 8.7% of SAD sufferers have sought medical treatment in Hong Kong (Lee et al., 2005), which means that most of the sufferers are undiagnosed and untreated. One of the most effective treatments for SAD is cognitive behavioral therapy (CBT), and internet-based CBT has shown promise in reducing general and social anxieties, as well as improving the quality of life of those with SAD (e.g. Carlbring et al., 2007; Tillfors et al., 2011). However, few studies have been conducted in this field in Hong Kong. This project aims to develop an online CBT program (including both an online platform and mobile application) for Hong Kong people with SAD, as well as evaluate its effectiveness in reducing anxiety symptoms and psychological distress, and improving quality of life at post-treatment and 3- and 6-month follow-ups. Randomized controlled trial (RCT) design was adopted for program evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents with fluency in Cantonese
* between the ages of 18 and 70
* a score of 25 or more on the Chinese version of the Social Phobia Inventory (C-SPIN) (Tsai et al., 2009)
* have not received any psychological treatment at the time of registration for participation in the project
* have access to a computer or smartphone with internet connection.

Exclusion Criteria:

* being severely depressed, with a score above 30 on the Beck Depression Inventory-II (BDI-II) (Beck, Steer & Brown, 1996)
* having suicidal ideation in the past three months, with a score of 3 points on Item 9 of the BDI-II.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Social Phobia Inventory | baseline: before the intervention program starts
  17-item rating scale for social anxiety symptoms, total scale score ratings from 0-68, with a higher score indicating a higher level of social anxiety.
Social Phobia Inventory | post-test: 1 month upon completion of the intervention program
  17-item rating scale for social anxiety symptoms, total scale score ratings from 0-68, with a higher score indicating a higher level of social anxiety.
Social Phobia Inventory | 3-month follow-up test: 3 months after completion of the intervention program
  17-item rating scale for social anxiety symptoms, total scale score ratings from 0-68, with a higher score indicating a higher level of social anxiety.
Social Phobia Inventory | 6-month follow-up test: 6 months after completion of the intervention program
  17-item rating scale for social anxiety symptoms, total scale score ratings from 0-68, with a higher score indicating a higher level of social anxiety.

SECONDARY OUTCOMES:
Beck Anxiety Inventory | baseline: before the intervention program starts
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Beck Anxiety Inventory | post-test: 1 month upon completion of the intervention program
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Beck Anxiety Inventory | 3-month follow-up test: 3 months after completion of the intervention program
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Beck Anxiety Inventory | 6-month follow-up test: 6 months after completion of the intervention program
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Beck Depression Inventory | baseline: before the intervention program starts
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptoms
Beck Depression Inventory | post-test: 1 month upon completion of the intervention program
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptoms
Beck Depression Inventory | 3-month follow-up test: 3 months after completion of the intervention program
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptoms
Beck Depression Inventory | 6-month follow-up test: 6 months after completion of the intervention program
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptoms
General Health Questionnaire-12 | baseline: before the intervention program starts
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
General Health Questionnaire-12 | post-test: 1 month upon completion of the intervention program
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
General Health Questionnaire-12 | 3-month follow-up test: 3 months after completion of the intervention program
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
General Health Questionnaire-12 | 6-month follow-up test: 6 months after completion of the intervention program
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
Automatic Thoughts Questionnaire | baseline: before the intervention program starts
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought.
Automatic Thoughts Questionnaire | post-test: 1 month upon completion of the intervention program
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought.
Automatic Thoughts Questionnaire | 3-month follow-up test: 3 months after completion of the intervention program
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought.
Automatic Thoughts Questionnaire | 6-month follow-up test: 6 months after completion of the intervention program
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought.
WHO Quality of life Scale-BREF | baseline: before the intervention program starts
  28-item rating scale for quality of life, including 2 items that measure the overall quality of life and 26 items that measure physical and psychological health, social relationships and the environment. Item score ranges from 1 (very dissatisfied) to 5 (very satisfied), with a higher score indicating better quality of life.
WHO Quality of life Scale-BREF | post-test: 1 month upon completion of the intervention program
  28-item rating scale for quality of life, including 2 items that measure the overall quality of life and 26 items that measure physical and psychological health, social relationships and the environment. Item score ranges from 1 (very dissatisfied) to 5 (very satisfied), with a higher score indicating better quality of life.
WHO Quality of life Scale-BREF | 3-month follow-up test: 3 months after completion of the intervention program
  28-item rating scale for quality of life, including 2 items that measure the overall quality of life and 26 items that measure physical and psychological health, social relationships and the environment. Item score ranges from 1 (very dissatisfied) to 5 (very satisfied), with a higher score indicating better quality of life.
WHO Quality of life Scale-BREF | 6-month follow-up test: 6 months after completion of the intervention program
  28-item rating scale for quality of life, including 2 items that measure the overall quality of life and 26 items that measure physical and psychological health, social relationships and the environment. Item score ranges from 1 (very dissatisfied) to 5 (very satisfied), with a higher score indicating better quality of life.
Internalized Stigma of Mental Illness | baseline: before the intervention program starts
  24-item rating scale for the subjective experiences of self-stigma on mental illness. It consists of 4 subscales: shame/alienation, stereotype endorsement, perceived discrimination and social withdrawal. Item score ranges from "1" ("strongly disagree") to "4" ("strongly agree"). All items are averaged as a scale score, with a higher score indicating a higher level of self-stigma.
Internalized Stigma of Mental Illness | post-test: 1 month upon completion of the intervention program
  24-item rating scale for the subjective experiences of self-stigma on mental illness. It consists of 4 subscales: shame/alienation, stereotype endorsement, perceived discrimination and social withdrawal. Item score ranges from "1" ("strongly disagree") to "4" ("strongly agree"). All items are averaged as a scale score, with a higher score indicating a higher level of self-stigma.
Internalized Stigma of Mental Illness | 3-month follow-up test: 3 months after completion of the intervention program
  24-item rating scale for the subjective experiences of self-stigma on mental illness. It consists of 4 subscales: shame/alienation, stereotype endorsement, perceived discrimination and social withdrawal. Item score ranges from "1" ("strongly disagree") to "4" ("strongly agree"). All items are averaged as a scale score, with a higher score indicating a higher level of self-stigma.
Internalized Stigma of Mental Illness | 6-month follow-up test: 6 months after completion of the intervention program
  24-item rating scale for the subjective experiences of self-stigma on mental illness. It consists of 4 subscales: shame/alienation, stereotype endorsement, perceived discrimination and social withdrawal. Item score ranges from "1" ("strongly disagree") to "4" ("strongly agree"). All items are averaged as a scale score, with a higher score indicating a higher level of self-stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayan Pan, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Jiayan Pan, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan JY. Internet-Based Cognitive Behavioral Therapy and Virtual Reality Exposure Therapy for Social Anxiety Disorder: Protocol for a Randomized Controlled Trial in Hong Kong. JMIR Res Protoc. 2023 Sep 14;12:e48437. doi: 10.2196/48437. PMID 37707944